CLINICAL TRIAL: NCT01867008
Title: Safety and Efficacy of the Cochlear Nucleus CI422 Cochlear Implant in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-CI422-2012
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Nucleus CI422 Cochlear Implant with Nucleus 6 (N6) Sound Processor (Experimental)
  Interventions: Device: Nucleus CI422 Cochlear Implant with N6 Sound Processor

INTERVENTIONS:
Device: Nucleus CI422 Cochlear Implant with N6 Sound Processor

SUMMARY:
Clinical study to evaluate the safety and efficacy of the Cochlear™ Nucleus® CI422 cochlear implant for new cochlear implant adult recipients with broader requirements to be considered an eligible candidate.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older at the time of implantation
2. Moderate low frequency thresholds up to and including 1000 Hz, severe to profound high frequency (above 3000 Hz) sensorineural hearing loss
3. Minimum of 30 days experience with appropriately fit bilateral amplification, fit using the standardized National Acoustics Laboratory (NAL) fitting method described in the Fitting and Use of Hearing Aids section below
4. Aided Consonant Nucleus Consonant (CNC) word recognition score (mean of two lists) between 10% and 50%, inclusive in the ear to be implanted
5. Aided CNC word recognition score (mean of two lists) in the contralateral ear equal to, or better than, the ear to be implanted but not more than 70%
6. Willingness to use bimodal stimulation (i.e., a cochlear implant on one ear and a hearing aid on the contralateral ear) through at least 6-months postactivation
7. English spoken as a primary language

Exclusion Criteria:

1. Duration of severe-to-profound hearing loss greater than 30 years
2. Congenital hearing loss (for the purpose of this study, onset prior to 2 years-of-age)
3. Medical or psychological conditions that contraindicate undergoing surgery as determined by the Investigator
4. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
5. Conductive overlay of 15 decibels (dB) or greater at two or more frequencies, in the range 500 to 1000 Hz
6. Deafness due to lesions of the acoustic nerve or central auditory pathway
7. Absence of cochlear development
8. Diagnosis of auditory neuropathy
9. Active middle-ear infection
10. Tympanic membrane perforation in the presence of active middle ear disease
11. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices as determined by the Investigator
12. Unwillingness or inability of the candidate to comply with all investigational requirements as determined by the Investigator
13. Additional handicaps that would prevent or restrict participation in the audiological evaluations as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Nucleus CI422 Cochlear Implant With N6 Sound Processor: Newly implanted patient population seeking cochlear implantation as standard of care
Period: Overall Study
Arm/Group | Nucleus CI422 Cochlear Implant With N6 Sound Processor
Started | 55
Completed | 54
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Nucleus CI422 Cochlear Implant With N6 Sound Processor: Newly implanted adults with moderate to severe sensorineural hearing loss, seeking cochlear implantation as a standard of care
Arm/Group | Nucleus CI422 Cochlear Implant With N6 Sound Processor
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Open Set Monosyllabic Word Recognition Score as Measured on a Consonant Nucleus Consonant (CNC) Word Test
Description: Performance at 6 months postactivation compared to pre-operative word recognition score (percent correct: 0-100%, where a 0% is the lowest score and a 100% is the highest score)
Time Frame: Preoperative baseline to 6 months postactivation
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | Nucleus CI422 Cochlear Implant With N6 Sound Processor
Number analyzed (Participants) | 54
percentage correct | 54.7 (21.3)

ADVERSE EVENTS:
Arm/Group | Nucleus CI422 Cochlear Implant With N6 Sound Processor
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 5/55
Other Adverse Events (participants affected / at risk) | 34/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus CI422 Cochlear Implant With N6 Sound Processor (N=55)
Irregular heartbeat (Cardiac disorders) | 1 (1) — Admitted overnight for irregular heartbeat
Broken hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo or dizziness (Ear and labyrinth disorders) | 1 (1) — Vertigo started 1 day post-op after discharged from surgery. Admitted for observation and provided steroids.
Atrial fibrillation (Cardiac disorders) | 1 (1) — Admitted to hospital for atrial fibrillation. Discharged without further episodes.
Revision surgery (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus CI422 Cochlear Implant With N6 Sound Processor (N=55)
New or worsened tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo or dizziness (Ear and labyrinth disorders) | 7 (7)
Skin flap (Ear and labyrinth disorders) | 1 (1)
Device related/programming problems (Ear and labyrinth disorders) | 5 (5)
Hearing loss (Ear and labyrinth disorders) | 9 (9)
Earmold or acoustic component sores (Ear and labyrinth disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-04-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT01867008/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT01867008/Prot_ICF_001.pdf